CLINICAL TRIAL: NCT02653066
Title: HealtheRx Survey for Pulmonary Research Registry Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-1282
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Asthma; COPD
Keywords: recruitment
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Participant is recruited via usual avenues including flyers and physician referral. This includes participants who received a HealtheRx with advertisement for phone survey but did not call in based on advertisement.
- Intervention with consent form (Experimental): After completing survey, participant in HealtheRx+ group receives $5 bill with their survey check and blank registry consent form.
  Interventions: Other: HealtheRx+
- Intervention with return of consent form (Experimental): After returning signed consent form, participant in HealtheRx++ group is mailed $5 bill.
  Interventions: Other: HealtheRx++

INTERVENTIONS:
Other: HealtheRx+ — Participant receives $5 bill with incentive check and blank consent form
  Arms: Intervention with consent form
Other: HealtheRx++ — Participant receives $5 bill when they returned signed PRR consent form.
  Arms: Intervention with return of consent form

SUMMARY:
The purpose of this research is to study the utility of using the HealtheRx as a tool to recruit eligible patients into the Pulmonary Research Registry (PRR) (IRB 15543B) at the University of Chicago. HealtheRx is an example of a potential recruitment tool that has high reach in populations typically underrepresented in research studies, uses a high tech infrastructure that allows matching of research opportunities to patient characteristics, but that delivers information in a low-tech, patient-centered mode using the printed HealtheRx prescription.

DETAILED DESCRIPTION:
1. Patients living in one of 16 zip codes of the South and West Sides of Chicago who present for care at one or more of 30 clinical sites receive a personalized HealtheRx prescription with programs and services in the community from their health care provider. The HealtheRx is printed and delivered to the patient at the end of the visit.
2. Patients age 18+ with a diagnosis of asthma and/or COPD will receive a HealtheRx with programs/services to help manage their condition, as well as an advertisement to participate in a phone survey.
3. Patients interested in completing the phone survey can call or text the Lindau Lab at the University of Chicago.
4. An experienced survey researcher will first read the consent script and if oral consent is received, continue with the phone survey (The survey includes items pertaining to program participants' receipt of the HealtheRx, use of community services provided on the HealtheRx, thoughts about participation in clinical research.
5. Participants who choose to complete the survey will receive a $10 check delivered via U.S. mail to their home address. Patients interested in joining the PRR will receive the PRR consent form with their $25 check.
6. Participants with interest in joining the PRR will also receive, via mail, a $5 bill as thanks for reading, signing and returning the consent form. Participants will be randomized to receive the $5 bill at 2 different time points.
7. Once the signed consent form is received, a member of the Asthma and COPD Center research staff will contact the participant by phone and complete the PRR case report form by phone.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of asthma/COPD
* receipt of HealtheRx

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Cost per consented subject | 6 months

SECONDARY OUTCOMES:
Mean number of consented subjects per week | 6 months

OTHER OUTCOMES:
Proportion of individuals who consent | 6 months
Mean days to consent | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Lindau, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Feldmeth G, Naureckas ET, Solway J, Lindau ST. Embedding research recruitment in a community resource e-prescribing system: lessons from an implementation study on Chicago's South Side. J Am Med Inform Assoc. 2019 Aug 1;26(8-9):840-846. doi: 10.1093/jamia/ocz059. PMID 31181137